CLINICAL TRIAL: NCT01605006
Title: HDE Post-Approval Study (PAS) of NeuRx DPS for ALS
Brief Title: Humanitarian Device Exemption Post-Approval Study of NeuRx Diaphragm Pacing System for Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 20-0009-0020
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: amyotrophic lateral sclerosis; ALS; motor neuron disease; diaphragm; diaphragm pacing; diaphragmatic pacing; phrenic pacing; phrenic nerve; phrenic nerve stimulation; NeuRx DPS; DPS; chronic hypoventilation; respiration; ventilation; breathing; Humanitarian Device Exemption; HDE; post-approval study
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NeuRx Diaphragm Pacing System (DPS) (Other): Surgical implantation of the NeuRx DPS (on label use).
  Interventions: Device: NeuRx Diaphragm Pacing System (DPS)

INTERVENTIONS:
Device: NeuRx Diaphragm Pacing System (DPS) — The NeuRx DPS is a percutaneous, intramuscular, diaphragm stimulation system which is implanted using standard laparoscopic surgical techniques in an outpatient procedure. The implanted intramuscular diaphragm electrodes are connected to a four channel external stimulator at a percutaneous exit site. DPS is designed to help ALS patients breathe by providing conditioning stimulation of the diaphragm muscles. Recommended frequency of diaphragm conditioning is at least 3 times per day with each session lasting at least 30 minutes. Patients may find it helpful to use the DPS for longer periods to help with breathing. DPS may be used at the same time as non-invasive ventilation. Patents may also sleep with the DPS to assist with breathing difficulties at night.
  Other Names: diaphragm pacing; diaphragmatic pacing; phrenic nerve stimulation

SUMMARY:
This post-approval study will follow 60 participants who have ALS, documented chronic hypoventilation, and bilateral phrenic nerve function, and who undergo the surgical implantation procedure to receive the NeuRx Diaphragm Pacing System device. Participants who are successfully implanted with the device will use it for daily diaphragm conditioning sessions. Participants will be followed for at least two years (until the last enrolled participant reaches the 2-year follow-up visit). Safety and probable benefit outcome measures will be assessed.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label, interventional, post-approval (FDA) study of the NeuRx Diaphragm Pacing System (DPS) device. The study will enroll 60 participants who have amyotrophic lateral sclerosis (ALS), meet the FDA-approved device indications for use, and undergo the surgical implantation procedure to receive the device. The device is intended for use in ALS patients with a stimulatable diaphragm (both right and left portions) as demonstrated by voluntary contraction or phrenic nerve conduction studies, and who are experiencing chronic hypoventilation (CH), but not progressed to an FVC less than 45% predicted. Participants who are successfully implanted with the device will use it for daily diaphragm conditioning sessions. Participants will be followed for at least two years (until the last enrolled participant reaches the 2-year follow-up visit). Safety and probable benefit outcome measures will be assessed. The primary objective of the study is: (1) (Safety) Characterize the types and frequency of major device-related adverse events (AEs) over the time of device use. Secondary objectives of the study are: (2) (Safety) Determine whether the frequency of major device-related AEs increases dramatically toward end of life; and (3) (Probable Benefit) Determine whether there is a relationship between survival time and onset type (bulbar and limb), time from onset to treatment, and use of NIV, riluzole, or PEG in patients treated with the device.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 or older.
2. Participants with familial or sporadic ALS diagnosed as laboratory-supported probable, probable, or definite according to the World Federation of Neurology El Escorial criteria.
3. Bilateral phrenic nerve function clinically acceptable as demonstrated by bilateral diaphragm movement with fluoroscopic sniff test or with EMG recordings and nerve conduction times.
4. Chronic hypoventilation was documented by at least one of the following:

   * FVC less than 50% predicted, or
   * |MIP| less than 60 cmH2O, or
   * PaCO2 greater than or equal to 45 mmHg, or
   * Nocturnal SaO2 less than or equal to 88% for at least five continuous minutes
5. Suitable surgical candidate.
6. Negative pregnancy test in female participants of childbearing potential.
7. Informed consent from patient or designated representative.

Exclusion Criteria:

1. Underlying cardiac or pulmonary disease that would increase the risk of general anesthesia.
2. Underlying pulmonary diseases that were present prior to ALS that would affect pulmonary tests independent of ALS.
3. Uncontrolled excessive secretions.
4. FVC less than 45% predicted at time of surgery.
5. Preexisting implanted electrical device such as pacemaker or cardiac defibrillator.
6. Pre-existing diaphragm abnormality such as a hiatal hernia or paraesophageal hernia of abdominal contents going into the thoracic cavity.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Safety Outcome Measure -- Occurrence of major device-related (including procedure-related) adverse events as defined below. | follow-up assessments at 3-month intervals
  * Serious capnothorax requiring invasive intervention
  * Mechanical ventilation for 24 hours or longer post-procedure
  * Post-procedure extubation failure resulting in permanent tracheostomy ventilation
  * Perioperative complication which delays initiation of NeuRx DPS therapy
  * Severe discomfort due to stimulation which is unable to be tolerated or resolved
  * Device malfunction which interrupts or causes an undesired diminution of NeuRx DPS therapy
  * Electrode dislodgement from the diaphragm
  * Wire infection
  * Any other device- or procedure-related serious adverse event

SECONDARY OUTCOMES:
Probable Benefit Outcome Measure | follow-up assessments at 3-month intervals
  Survival, defined as time to (a) death or (b) permanent tracheostomy mechanical ventilation (PTV) with discontinuation of pacing. (All deaths and PTV events will be reported regardless of relationship to the device or procedure.)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Miller, M.D., Principal Investigator — Forbes Norris MDA/ALS Research Center, California Pacific Medical Center
Locations (11):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center -- Forbes Norris MDA/ALS Research Center, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Stony Brook University, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Summary of Safety and Probable Benefit for Humanitarian Device Exemption (Approved September 28, 2011) — http://www.accessdata.fda.gov/cdrh_docs/pdf10/H100006b.pdf